CLINICAL TRIAL: NCT00364728
Title: Efferocytosis (Clearance of Apoptotic Cells by Phagocytosis) and Autoimmune Diseases in Human
Brief Title: Efferocytosis and Genomic Polymorphism in Autoimmune Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: National Taiwan University Hospital research ethics committee, National Taiwan University Hospital
Other Study IDs: 9561701025; NSC98-2320-B-002-021-MY2
Record Dates: First submitted 2006-08-15; First posted 2006-08-16 (Estimated); Last update posted 2010-05-21 (Estimated); Status verified 2010-05

CONDITIONS: SLE; Rheumatoid Arthritis; Healthy Subjects
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Over the past few years, growing evidences revealed that clearance of apoptotic cells by phagocytosis can result in powerful anti-inflammatory and immunosuppressive effects. In vivo, apoptotic cells are cleared rapidly by neighboring cells, macrophages and related scavengers. Defective clearance of apoptotic cells has been linked closely to autoimmunity and persistent inflammatory disease. Several phagocytic receptors, bridging molecules produced by phagocytes and 'eat-me' signals on apoptotic cells are coordinately involved in mediating clearance of apoptotic cells. Complement receptors (CR3, CR4), collection, CD14, CD36 (Class B scavenger receptor), class A scavenger receptor, asialoprotein receptor, Mer receptor kinase were reported to recognize apoptotic cells. The best characterized system for clearance of apoptotic cells is the recognition of phosphatidylserine (PS) on apoptotic cells by phosphatidylserine receptor (PSR). Milk fat globule- epidermal growth factor 8 (MFG-E8) is an opsonin that bridges phagocytes (by interacting with α vβ3, αvβ5 integrins via RGD motif) and apoptotic cells (by binding PS through Factor V/VIII-C domain). Activated macrophages produce and secret MFG-E8. MFG-E8 is a critical component in PSR-mediated phagocytosis of apoptotic cells. The dominant negative mutant MFG-E8, D89E, that carried a mutated RGD motif inhibited phagocytosis of apoptotic cells in vitro. Injection of D89E into wild type mice induced autoantibodies and IgG deposition on glomeruli. Macrophages from MFG-E8 deficiency (MFG-E8-/-) mice were impaired in engulfment of apoptotic cells, which can be restored by adding recombinant MFG-E8. The female MFG-E8-/- mice spontaneously produced high titer of autoantibodies and developed lupus-like glomerulonephritis at the age of week 40. Defective clearance of apoptotic cells is closely related to development of autoimmunity. In the past 4 years, a growing number of molecules were recognized as receptors for the PS exposed on the apoptotic cells. These molecules were capable of mediating phagocytic clearance, rendering anti-inflammatory cytokines in the phagocytes, and modulating T cell responses.

The specific aim of this proposal is to study genetic polymorphism in MFG-E8, PSR and other factors implicated in phagocytic clearance of apoptotic cells among Taiwanese. By comparing the polymorphism between patients with autoimmune disease (SLE or RA) and healthy control subjects, we will investigate if genetic variations among individuals of genes encoding proteins involved in clearance of apoptotic cells contribute to the pathogenesis of systemic autoimmune diseases SLE and RA.

DETAILED DESCRIPTION:
Over the past few years, there were growing evidences that clearance of apoptotic cells by phagocytosis can result in powerful anti-inflammatory and immunosuppressive effects. The defective clearance of apoptotic cells has been linked to autoimmunity and persistent inflammatory diseases. Apoptotic cells are cleared in vivo rapidly. Clearance of apoptotic cells or apoptotic bodies is histologically undetectable in normal situation by neighboring cells, or by macrophages and related scavengers. Defective clearance of apoptotic cells has been linked closely to autoimmune and persistent inflammatory diseases.

The process of discriminating apoptotic from live cells was found to be remarked complex. Many phagocytic receptors, bridging molecules, and several 'eat-me' markers on apoptotic cells are involved and coordinated interact with each other. A phagocytic-synapse interprets the apoptotic-cell-associated molecular pattern (ACAMPS), and determine the behaviors subsequent to phagocytosis.

Clearance of apoptotic cells can be mediated by complement receptors CR3 (CD116/CD18), CR4 (CD11c/CD18), collections and CD14. However, the clearance of apoptotic cells does not usually trigger either inflammation or an adaptive immune response. Clearance of apoptotic cells can also be mediated by receptors that were firstly characterized to clear damaged cells or altered-self-components.

The best characterized system for clearing the apoptotic cells is the recognition of phosphatidylerine on the apoptotic cells. Phosphatidylserine (PS) was found to distribute in the inner layer of plasma membrane phospholipid bi-layer in healthy cells. During apoptotic process, inhibition of aminophopholipid translocase and activation of lipid scramblase result in exposure of PS on the cell surface.

Defective macrophage clearance of apoptotic cells linked to autoimmunity. There were emerging evidences indicating defective macrophage clearance of apoptotic cells linked to autoimmunity.

1. Systemic exposure to irradiated apoptotic cells induces autoantibody production. Normal mice injected with 10^7 syngenic, apoptotic thymocytes developed transient and low titer of anti-nuclear antibody, anti-cardiolipin, and anti-ssDNA antibody. All immunized mice had IgG deposition in the glomeruli several months after immunization. IgG-deposition was not found in the glomeruli of non-immunized or syngenic splenocyte-immunized controls.
2. Defective clearance of apoptotic cells and SLE-like autoimmunity was found to be associated C1q deficiency. C1q mice developed systemic autoimmunity spontaneously, with a marked excess of free, non-ingested apoptotic cells of the kidney. Although congenital deficiency of complement cascade is rare in humans, nearly all patients who were deficient in C1q developed SLE-like disease. In both human and mice, inflammatory macrophages had defect in the uptake of apoptotic cells and the defect could be rescued by adding exogenous C1q.
3. Mer/kd (Mer knock-down) mice developed autoimmune disease Mer is a member of Ax1/Mer/Tyro3 receptor tyrosine kinase family. Growth arrest-specific gene 6 (GAS6) was shown to bridge Mer to phosphatidylserine on apoptotic cells. Mer-kd mice had macrophages deficient in clearance of apoptotic thymocytes. The phagocytic deficiency was restricted to apoptotic cells and was independent of Fc receptor-mediated phagocytosis or ingestion of other particles. Mer-kd mice developed progressive lupus-like immunity, with antibodies to chromatin, DNA, and IgG. The autoimmunity appears to be spontaneously, driven by endogenous antigens, with little polyclonal B cell activation.
4. Impaired phagocytosis of apoptotic material by monocyte-derived macrophages from patients with SLE. Reduced clearance of apoptotic cells in SLE patients was observed, although apoptosis was normally happened.

Milk fat globule-EGF factor 8 (MFG-E8) was characterized in mouse milk glycoproteins, 53 and 66 kD, peripherally associated with the membrane surrounding the lipid droplet (milk fat globule membrane, MFGM). MFG-E8 is expressed abundantly in lactating mammary glands and secreted in associated with milk fat globules.

MFG-E8 consists of two repeated EGF-like domains on the terminal side and tandem discoidin-like (C-) domains homologous to the C1 and C2 domains of coagulation factor V and VIII. The C2 domain can mediate Ca2+-independent binding to PS. MFG-E8 expression is up-regulated in lactating mammary gland, and has been detected in other tissues such as brain, lung, heart, kidney and spleen in mouse, bovine and human.

The second EGF-like domain of MFG-E8 contains an integrin-binding motif, namely Arg-Gly-ASP (RGD) sequence. The RGD motif is conserved in all known MFG-E8 sequence in different species. It can bind to αvβ3 and αvβ5 integrins. MFG-E8 was characterized as a peripheral membrane protein, although there was no apparent hydrophobic transmembrane domain, and bind directly to MFGM or cell membrane. The MFG-E8 binds to anionic phospholipids, especially phosphatidylserine, on the second C (C2) domain independent of Calcium ions.

Reports indicated that MFG-E8 secreted extracellularly despite its membrane associated nature. MFG-E8 was found to be a major component of secretory membrane vesicles (exosomes) secreted by murine dendric cell line, D1. The glioma cell line (C6) secrets MFG-E8 into the culture media. MFG-E8 is also detected in embryonic gonad extracellularly and in the sera of patients with metastatic tumor.

MFG-E8 was regards as an opsonin that bridge apoptotic cells, which with surface phoshatidylserine exposure, and phagocyte bearing αvβ3 and αvβ5 integrins. Hanayana et. al. showed that thioglycollate-elicited macrophages produced and secreted MFG-E8. MFG-E8 significantly bound to apoptotic cells by recognizing aminophospholipids such as phosphatidylserine and bound to macrophages via its RGD motif, particularly strongly to αvβ3 integrin. Transfected NIH3T3 cell with high αvβ5 expression can engulf apoptotic cell in the presence of MFG-E8. The MFG-E8 dominant negative mutant that carries a point mutation in the RGD motif inhibited phagocytosis of apoptotic cells by peritoneal macrophages in vivo and in vitro. Borisenko et. al. estimated that MFG-E8 bind 2~8 fold stronger to oxidized PS than to native PS. And they also proposed MFG-E8 might bind to another cofactor, annexin I, on apoptotic cells, thus increase protein-membrane interaction.

Human MFG-E8 gene was located on chromosome 15q25. The cDNA clone contains coding sequence for 387 ammo-acid peptides of which 263 (68%) are identical with mouse protein.

Tingible body macrophages, characterized by CD68+ F4/80-, in spleen and lymph node express significant level of MFG-E8. Peritoneal macrophages elicited by thioglycollate secrete abundant MFG-E8 protein of 74 kD in the culture supernatant. The macrophages from MFG-E8(-/-) mice engulf few apoptotic cells compared to the macrophages from their normal littermates in vitro. Addition of recombinant MFG-E8 in the culture restored the ability of MFG-E8(-/-) Mφs to engulf apoptotic cells in a doze-dependent manner.

In germinal centers, somatic hypermutation and secondary BCR rearrangement are involved in BCR affinity maturation. The modified BCRs with lower affinity will be removed by apoptosis. Tingible body macrophages are responsible for the MFG-E8-dependent clearance of apoptotic cells. Tingible body Mφs in wild type mice engulfed and digested the apoptotic B cells efficiently, whereas the MFG-E8(-/-) Mφs just wrapped many apoptotic cells without engulfment42. The MFG-E8(-/-) mice developed splenomegaly in an age-dependent manner. The white pulps in the spleens of the MFG-E8(-/-) mice were greatly enlarged and carried numerous germinal centers.

The follicular zones were enlarged. There were 2 to 3 times more lymphocytes in the spleens of the MFG-E8(-/-) mice. An increased number of IgG-producing cells were found in the spleen follicles. The female MFG-E8(-/-) mice spontaneously produced high titer of anti-antibodies anti-dsDNA and ANA at the age of week 40 but not at w10. Immunization female 10-week-old mice twice with KLH promoted ANA production 20 days later in MFG-E8(-/-) but not wild type mice. Immune complex deposition, hyper-cellularity of glomeruli, and proteinuria were observed in most female MFG-E8(-/-) mice at week 40. Therefore, inefficient engulfment of apoptotic B cells by might lead to lupus-like autoimmune disease. Kenichi et al. showed that masking phosphatidylserine by MFG-E8 mutant D89E, carrying a point mutation in RGD motif, inhibited not only the phagocytosis of apoptotic cells by macrophages of different origins but also the production of IL10 by thioglycollate-elicited peritoneal macrophages after phagocytosing apoptotic cells. When D89E MFG-E8 was injected into wild type mice intravenously, auto-antibodies were induced. The production of auto-antibodies was enhanced by co-injection of syngenic apoptotic cells. The auto-antibodies persisted for a long-term and IgG deposition on glomeruli took place. These results added in proof that the impairment of phagocytic clearance of apoptotic cells leads to auto-antibody production and autoimmune disease.In the past 4 years, a growing number of molecules were recognized as receptors for the PS exposed on the apoptotic cells. These molecules were capable of mediating phagocytic clearance, rendering anti-inflammatory cytokines in the phagocytes, and modulating T cell responses.

The specific aim of this proposal is to study genetic polymorphism in MFG-E8, PSR and other factors implicated in phagocytic clearance of apoptotic cells among Taiwanese. By comparing the polymorphism between patients with autoimmune disease (SLE or RA) and healthy control subjects, we will investigate if genetic variations among individuals of genes encoding proteins involved in clearance of apoptotic cells contribute to the pathogenesis of systemic autoimmune diseases SLE and RA.

Specific aim:

As described in the above introduction, in order to test if factors involved in clearance of apoptotic cells are implicated in pathogenesis of human autoimmune diseases, we intend to investigate if the genetic variation among individuals of genes encoding proteins involved in clearance of apoptotic cells, MFG-E8 and PSR, contributes to pathogenesis of human autoimmune diseases SLE and RA.

The goal of this proposal:

We will

1. Find out genetic polymorphism of human PSR gene in Taiwan by study single nucleotide polymorphism (SNPs) of PSR genes among Taiwanese subjects using PCR and DNA sequencing.
2. Study the PSR SNPs in SLE and RA patients and non-auto-immune control subjects by PCR/sequence-specific oligonucleotide probe hybridization.
3. Compare the allelic distribution of each SNP among patients and control group and find if there is disease-associated SNP(s) in PSR gene.
4. Find out genetic polymorphism of human MFG-E8 gene in Taiwan by study SNPs of MFG-E8 genes among Taiwanese subjects using PCR and DNA sequencing.
5. Study the MFG-E8 SNPs in SLE and RA patients and non-auto-immune control subjects by PCR/sequence-specific oligonucleotide probe hybridization.
6. Compare the allelic distribution of each SNP among patients and control group and find if there is disease-associated SNP(s) in MFG-E8 gene.

ELIGIBILITY:
Inclusion Criteria:

* SLE, RA, healthy

Exclusion Criteria:

* nil

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Taiwan autoimmune diseases case control study
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2006-01; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Yi Hu, PhD, Principal Investigator — Department of Clinical Laboratory Sciences and Medical Biotechnology
Locations (1):
- Chung-Yi Hu, Taipei, Taiwan, Taiwan